CLINICAL TRIAL: NCT01854099
Title: Peptide Targets for Glioblastoma Against Novel Cytomegalovirus Antigens
Brief Title: Peptide Vaccine for Glioblastoma Against Cytomegalovirus Antigens
Acronym: PERFORMANCE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator decided not to open study.
Sponsor: University of Florida (Other)
Collaborators: American Brain Tumor Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERFORMANCE
Record Dates: First submitted 2013-05-11; First posted 2013-05-15 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Glioblastoma
Keywords: Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 Day TMZ with PEP-CMV on Day 6-8 (Active Comparator): Standard TMZ (200 mg/m2/day x 5 days) with PEP-CMV vaccination on Day 6-8 of each monthly TMZ cycle
  Interventions: Biological: PEP-CMV
- 5 day TMZ with vaccine on day 22-24 (Active Comparator): Standard TMZ (200 mg/m2/day x 5 days) with vaccination on Day 22-24 of each monthly TMZ cycle
  Interventions: Biological: PEP-CMV
- 21 day TMZ wtih vaccine on day 22-24 (Active Comparator): Dose-intensified TMZ (100 mg/m2/day x 21 days) with vaccination on day 22-24 of each monthly TMZ cycle
  Interventions: Biological: PEP-CMV

INTERVENTIONS:
Biological: PEP-CMV — 500 µg of PEP-CMV vaccine given intradermally on day 6-8 of each monthly TMZ cycle (standard 200 mg/m^2 x 5 days) with group 1.
  Arms: 5 Day TMZ with PEP-CMV on Day 6-8
Biological: PEP-CMV — 500 µg of PEP-CMV vaccine given intradermally on day 22-24 of each monthly TMZ cycle (standard 200 mg/m^2 x 5 days) with group 2.
  Arms: 5 day TMZ with vaccine on day 22-24
Biological: PEP-CMV — 500 µg of PEP-CMV vaccine given intradermally on day 22-24 of each monthly TMZ cycle (dose-intensified 100 mg/m^2 x 21 days) with group 3.
  Arms: 21 day TMZ wtih vaccine on day 22-24

SUMMARY:
Eligible adult patients with new diagnosis of gliobastoma are enrolled to receive 3 weekly vaccinations of the study drug PEP-CMV 1-3 days following standard of care chemoradiation. Patients will then be randomized to one of three arms: 1). standard temozolomide (TMZ)(200mg/m^2 for 5 days) with vaccine on day 6-8 of each monthly TMZ cycle. 2). standard TMZ (200mg/m^2 for 5 days) with vaccine on day 22-24 of each monthly TMZ cycle. 3). dose-intensified TMZ (100 mg./m^2 for 21 days) with vaccine on day 22-24 of each monthly cycle. All vaccines will be given intradermally (i.d.) and will be given with monthly TMZ cycles and continue after TMZ cycles until progression or death.

DETAILED DESCRIPTION:
Eligible patients will be screened and enrolled prior to completion of post-surgical chemoradiation. Final eligibility to remain on study for safety endpoint will occur after completion of chemoradiation and prior to initiation of adjuvant TMZ regimen. Immediately post-chemoradiation and prior to initiation of cycle 1 of adjuvant TMZ, all patients will receive 500 µg of PEP-CMV vaccine weekly for a total of 3 vaccines starting 1-3 days after chemoradiation is complete. Prior to initiation of TMZ cycle 1, patients will be randomized to one of three arms (1:1:1) to receive (1) standard TMZ (200 mg/m^2/day x 5 days) with vaccination on Day 6-8 of each monthly TMZ cycle, (2) standard TMZ (200 mg/m^2/day x 5 days) with vaccination on Day 22-24 of each monthly TMZ cycle, or (3) dose-intensified TMZ (100 mg/m^2/day x 21 days) with vaccination on day 22-24 of each monthly TMZ cycle. Each cohort will have 20 patients. Up to 150 patients will be consented in order to obtain 60 evaluable patients.

The primary safety assessment for dose-limiting toxicity (DLT) will be determined one week after the third weekly vaccine. A DLT will be defined as any irreversible Grade 3 toxicity, any Grade 4 toxicity, or any life threatening-event not attributable to concomitant medication, co-morbid event, or disease progression. Initially 6 patients will be accrued to the study (2 per arm) after which accrual will be suspended to review the toxicity experienced by these patients during the first 3 weekly vaccinations. If 0 or 1 of these patients experience DLT, accrual of the remaining patients will commence. Otherwise, modifications of the protocol will be considered before accruing additional patients.

The prevalence of DLT occurring during the initial 3 weekly vaccinations or the vaccinations administered concurrently with temozolomide will be continuously monitored. If more than 25% of accrued patients experience DLT, then accrual will be suspended and reported toxicity will be carefully reviewed to determine if modifications to the protocol treatment should occur. Peptide vaccinations employing GM-CSF and Montanide ISA-51 as adjuvants have generally been well tolerated in human patients in numerous phase I-III trials.

Treatment Plan: One week after the 3rd weekly vaccination, cycles of TMZ will begin. The start of all subsequent cycles will be scheduled every 4 weeks after the first daily dose of the preceding cycle. During monthly TMZ cycles, vaccinations will occur on day 6-8 or day 22-24 of each cycle, depending on randomization arm. All vaccines will be given i.d. approximately 10cm below the inguinal ligament bilaterally. A target of six cycles with maximum of twelve cycles of TMZ may be given if the patient demonstrates continued improvement on MRI scan, decreased corticosteroid requirement, improvement in performance status, or improvement in neurologic function at the discretion of the treating neuro-oncologist. Vaccines will continue monthly after TMZ cycles until tumor progression or death.

Patients will be imaged with contrast-enhanced MRI pre & post-surgical resection (prior to initiation of chemoradiation), post-chemoradiation and prior to TMZ cycle 1, prior to TMZ cycle 4, 7 (if administered), and 10 (if administered). MRI imaging every 3 months during post-chemoradiation is preferable, but every 2 months is allowed at the discretion of the treating neuro-oncologist. MRI imaging will be conducted every 3 months after completion of TMZ for 1 year, and then every 6 months thereafter, or at frequency indicated by clinical presentation. The modified Response Assessment in Neuro-Oncology (RANO) criteria will be used for assessment of pseudoprogression and patients demonstrating definitive progression will be removed from study. Any patient removed for definitive tumor progression prior to receiving third vaccine and post vaccination immune monitoring blood draw will be replaced for safety and immunologic endpoints. Clinical endpoint comparisons will be made amongst patients successfully randomized to adjuvant TMZ treatment arms.

Blood for immune monitoring will be obtained prior to vaccines 1-4, 7 and 13, and at tumor progression. Patients seen by the Duke neuro-oncology team between these vaccine visits may have blood drawn for immune monitoring at the discretion of the study team.

As part of standard care for these patients, upon tumor progression, participants may undergo stereotactic biopsy or resection. As this is not a research procedure, consent will be obtained separately. Patients that have this procedure done here at Duke University Health System, may be approached to participate in the Duke Brain Tumor Center Biorepository study. Tissue obtained from patients who consented to the Duke Brain Tumor Center Biorepository will be used to assess immunologic cell infiltration, antigen expression, and biomarkers for immunologic response.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histopathologically proven newly-diagnosed primary glioblastoma multiforme.
* The tumor must have a supratentorial component.
* Patients must be CMV seropositive.
* Signed informed consent. If the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the responsible family member or legal representative.
* For females of child-bearing potential, negative serum pregnancy test 48 hours prior to temozolomide.
* Women of childbearing potential and male participants must practice adequate contraception.
* Karnofsky performance status of ≥ 60.
* Patients must have recovered from the effects of surgery, postoperative infection, and other complications at time of enrollment.

Prior to adjuvant TMZ:

* Patients must complete radiation therapy (RT) (60.0Gy over 6 weeks) and concomitant TMZ (targeted dose of 75mg/m2/d for <49 days) therapy without significant toxicity that persisted over a duration of 4 weeks. Significant toxicity is defined as one or more of the following observations:

  * Absolute neutrophil count (ANC) < 0.5 x 109/L (Grade 4)
  * Platelet count < 10 x 109/L (Grade 4)
  * Grade 3 or 4 non-hematologic adverse event (AE) (except alopecia, nausea and vomiting unless the patient has failed maximal antiemetic therapy, and fatigue).
* Documentation of stable or decreasing steroid dose prior to randomization with goal of minimizing steroid use.
* CBC/differential with adequate bone marrow function as defined below:

  1. ANC, ≥ 1500 cells/mm^3. Platelet count, ≥ 100,000 cells/mm^3.
  2. Hemoglobin ≥ 10 g/dl. (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10 g/dl is acceptable.)
* Adequate renal function prior to vaccination as defined below:

  a. Blood Urea Nitrogen (BUN) ≤ 25 mg/dl Creatinine ≤ 1.7 mg/dl
* Adequate hepatic function prior to vaccination as defined below:

  1. Bilirubin ≤ 2.0 mg/dl
  2. ALT ≤ 3 x normal range
  3. AST ≤ 3 x normal range

Exclusion Criteria:

* Patients did not start RT and TMZ within 5 weeks of surgery.
* Patients that did not complete 60.0Gy over 6-7 weeks of RT (patients consented prior to completion who do not complete RT will be removed from study and replaced).
* Progression of disease prior to randomization as defined by RANO.
* Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years. (For example, carcinoma in situ of the breast, oral cavity, and cervix are all permissible.)
* Metastases detected below the tentorium or beyond the cranial vault.
* Prior chemotherapy or radiosensitizers (including Gliadel wafers) for cancers of the head and neck region (other than TMZ prescribed during radiation for glioblastoma); note that prior chemotherapy for a different cancer is allowable.
* Prior radiotherapy to the head or neck (except for T1 glottic cancer and that prescribed for GBM ≤60 Gy), resulting in overlap of radiation fields. Radiosurgery is not permitted.
* Severe, active co-morbidity, defined as follows:

  1. Unstable angina and/or congestive heart failure requiring hospitalization.
  2. Transmural myocardial infarction within the last 6 months.
  3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of beginning chemoradiation.
  4. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of beginning chemoradiation.
  5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
  6. Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
  7. Major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
  8. Active connective tissue disorders, such as lupus or scleroderma that in the opinion of the treating physician may put the patient at high risk for radiation toxicity.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
* Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant due to study drug.
* Prior allergic reaction to temozolomide or Keyhole Limpet Hemocyanin (KLH).
* Patients treated on any other therapeutic clinical protocols within 30 days prior to study entry or during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months
  To determine the optimal & safe peptide vaccination regimen with TMZ through dose-limiting toxicity (DLT) measurements. The primary safety assessment for DLT will be determined 1 week after the 3rd weekly vaccine. A DLT will be defined as any irreversible Grade 3 toxicity, any Grade 4 toxicity, or any life threatening-event not attributable to concomitant medication, co-morbid event, or disease progression. Initially 6 patients will be accrued to the study (2 per arm) after which accrual will be suspended to review the toxicity experienced by these patients during the first 3 weekly vaccinations. If 0 or 1 of these patients experience DLT, accrual of the remaining patients will commence. Otherwise, modifications of the protocol will be considered before accruing additional patients.

CONTACTS AND LOCATIONS:
Overall Officials: Duane A Mitchell, MD, PhD, Principal Investigator — University of Florida